CLINICAL TRIAL: NCT05567068
Title: Repurposing Atorvastatin in Patients With Ulcerative Colitis Treated With Mesalamine by Modulation of mTOR/NLRP3 Pathway.
Brief Title: Atorvastatin Efficacy and Safety in Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Bahaa, Teaching Assistant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3433
Record Dates: First submitted 2022-10-01; First posted 2022-10-05 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Atorvastatin; Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: double-blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): This group will take mesalamine 1 g three times daily
  Interventions: Drug: Mesalamine
- Atorvastatin group (Active Comparator): This group will take mesalamine 1 g three times daily plus atorvastatin 80 mg once daily.
  Interventions: Drug: Atorvastatin 80mg; Drug: Mesalamine

INTERVENTIONS:
Drug: Atorvastatin 80mg — Atrovastatin is one of the most effective drugs used to reduce intracellular cholesterol synthesis. it exerts numerous pleiotropic effects including anti-inflammatory, antioxidant properties, endothelial function improvement and immunomodulation independent of its basic lipid-lowering properties
  Arms: Atorvastatin group
Drug: Mesalamine — Mesalamine

SUMMARY:
Statins exert numerous pleiotropic effects including anti-inflammatory, antioxidant properties, endothelial function improvement, and immunomodulation independent of their basic lipid-lowering properties.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Both males and females will be included
* Negative pregnancy test and effective contraception.

Exclusion Criteria:

* Breastfeeding
* Significant liver and kidney function abnormalities
* Colorectal cancer patients
* Patients with severe UC
* Patients taking rectal or systemic steroids
* Patients taking immunosuppressives or biological therapies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Improvement in health related quality of life | 6 months
  HRQL questionnaire will be assessed according to bowel symptoms, emotional symptoms, systemic symptoms, and social symptoms

SECONDARY OUTCOMES:
changes in serum and fecal inflammatory biomarkers | 6 months
  The secondary endpoint is estimated by changes in serum IL-18, and fecal calprotectin.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Derived] Khrieba MO, Abdulelah FM, Alsaleh NA, AlRasheed HA, Ahmed TI, El-Sayed Mansy A, Hamouda MA, Habba E, Elshorbagi N, Abd Elhameed AG, Hamza E, Salahuddin MM, Mourad SA, Kamal M. Atorvastatin as an immunomodulatory adjunct in ulcerative colitis, beyond lipid lowering to inflammation control: a randomized controlled pilot study. Front Pharmacol. 2025 Oct 29;16:1690513. doi: 10.3389/fphar.2025.1690513. eCollection 2025. PMID 41235106